CLINICAL TRIAL: NCT03193294
Title: CORonary MICrovascular Angina (CorMicA): a Randomised, Controlled, Pilot Trial
Brief Title: CORonary MICrovascular Angina (CorMicA)
Acronym: CorMicA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NHS National Waiting Times Centre Board (Other)
Collaborators: British Heart Foundation (Other)
Responsible Party: Principal Investigator, Colin Berry, Professor of Cardiology and Imaging, NHS National Waiting Times Centre Board
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 16CARD25
Record Dates: First submitted 2017-06-13; First posted 2017-06-20 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Angina, Stable; Coronary Vasospasm; Coronary Circulation; Coronary Syndrome; Microvascular Angina; Coronary Disease
MeSH Terms: conditions — Angina, Stable; Coronary Vasospasm; Angina, Unstable; Microvascular Angina; Coronary Disease

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, parallel group, prospective
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants are randomised to a 'Disclosed group' (Intervention group) or a 'Not disclosed group' (Standard Care). In the standard care group, coronary function parameters are measured but the results are not disclosed to the attending clinician or the participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (coronary function test results disclosed) (Active Comparator): In the intervention group, coronary function tests are measured and disclosed to the attending clinician permitting re-evaluation of the initial diagnosis and treatment as compared with initial angiography-guided decisions. The intervention involves measurement of CFR, IMR and RRR in a target, major coronary artery followed by coronary reactivity testing using incremental doses of acetylcholine (10-4M, 10-5M, 10-6M) to assess endothelial function, bolus infusion of ACh (10-4M) for vasospasm provocation testing, followed by administration of a bolus dose (300 micrograms) of glyceryl trinitrate. Endotypes are identified based on established criteria for abnormalities in coronary vasodilator function, vasospasm and microvascular resistance. The endotypes (diagnostic strata) are: obstructive CAD, coronary artery spasm, microvascular angina, endothelial dysfunction (no angina), normal (non-cardiac). A diagnosis may be ruled-in or ruled-out based on the test results.
  Interventions: Diagnostic Test: Stratified medicine involving a diagnostic intervention
- Usual care group (coronary function results not disclosed) (Sham Comparator): Coronary function tests are measured but not disclosed to the attending clinician or the participant. The same coronary function tests are undertaken as in the intervention group. Masking is achieved by obscuring the catheter laboratory monitors from the attending clinician and participant. The effectiveness of masking is prospectively monitored.
  Interventions: Diagnostic Test: Stratified medicine involving a diagnostic intervention

INTERVENTIONS:
Diagnostic Test: Stratified medicine involving a diagnostic intervention — Adjunctive tests of coronary artery function at the time of invasive coronary angiography. Diagnostic groups: stable coronary syndromes in patients with no-obstructive coronary artery disease including the following sub-groups (coronary artery vasospasm, microvascular spasm, impaired vasorelaxation due to (1) endothelial dysfunction and/or (2) non-endothelial dysfunction, or unaffected (normal test results). Medical management is linked to contemporary clinical guidelines for the management of patients with stable coronary artery disease (European Society of Cardiology (2013)).

SUMMARY:
Angina is form of chest pain that is due to a lack of blood to the heart muscle. Angina is commonly triggered by stress and exertion, and is a common health problem worldwide. The diagnosis and treatment of angina is usually focused on detection of blockages in heart arteries, and relief of this problem with drugs, stents or bypass surgery. However, about one third of all invasive angiograms that are performed in patients with angina do not reveal any blockages. Many of such patients may have symptoms due to narrowings in the very small micro vessels (too small to be seen on an angiogram). The purpose of this research is to undertake a 'proof-of-concept' clinical trial to gather information as to whether routine tests of small vessel function in the heart might help identify patients with a stable coronary syndrome due to a disorder of coronary function (vasospastic or microvascular angina), and appropriately rule out this problem in patients with normal test results. The diagnostic strategy enables stratification of patient sub-groups to optimized therapy (personalised medicine). Evidence of patient benefits in this study would support the plan for a larger study that would be designed to impact on healthcare costs and patient reported outcome measures (PROMS).

DETAILED DESCRIPTION:
Background: Patients with a stable coronary syndromes include those with obstructive coronary artery disease (CAD) or ischaemia with no obstructive CAD (INOCA). Disorders of coronary vasomotion leading to microvascular and vasospastic angina are debilitating, prognostically important health problems. Use of coronary function tests with thresholds (normal/abnormal) that are linked to evidence-based treatment (start/stop) could be useful to diagnose (rule-in/rule-out) these conditions, but, evidence is lacking.

Design: (1) A proof-of-concept, randomised controlled stratified medicine trial of a clinical strategy informed by invasive tests of coronary function and linked guideline-based treatment decisions vs. standard care using angiography only in 150 patients; (2) A nested observational imaging sub-study using quantitative stress perfusion cardiac magnetic resonance (CMR). CONSORT guidelines will be followed.

Objectives: (1) To assess whether a diagnostic strategy involving tests of coronary function changes the diagnosis and treatment and improves health and economic outcomes; (2) To assess the diagnostic accuracy of novel MRI methods for abnormal perfusion due to microvascular disease.

Methods: Patients undergoing invasive coronary angiography for the investigation of known or suspected angina and who do not have either structural heart disease or a systemic health problem that would explain those symptoms will be invited to participate. Written informed consent is required for participation. Eligibility is further confirmed at the time of the coronary angiogram by exclusion of obstructive (>50% stenosis, fractional flow reserve <=0.80) coronary artery disease (CAD). After the angiogram, eligible participants will be randomised immediately in the catheter laboratory to test disclosure (intervention group) or measurement without disclosure (control group). Coronary function will be assessed using a diagnostic guidewire and intra-coronary infusions of acetylcholine (10-6M, 10-5M, -10-4M) and a bolus of glyceryl trinitrate (300 micrograms). The guidewire-derived parameters include fractional flow reserve (FFR), coronary flow reserve (CFR), index of microvascular resistance (IMR) and the resistance reserve ratio (RRR). Participants who are enrolled but not randomised will enter a follow-up registry. The endotypes (diagnostic strata) are: obstructive CAD, coronary vasospastic angina, microvascular angina, endothelial dysfunction (no angina), normal (non-cardiac, normal coronary function results, no angina). Thus, a diagnosis may be ruled-in or ruled-out based on the test results. Microvascular disease will be characterised as structural (abnormal IMR) and/or functional (abnormal CFR, RRR). Primary outcome: Between-group difference in Seattle Angina Questionnaire (SAQ) scores at 6 months; Secondary: Reclassification of the treatment decision; certainty of the diagnosis; health status (EQ-5D, Illness Perception, Treatment Satisfaction & Patient Health questionnaires); angina medication and adherence; health economics; reference clinical decisions as evaluated by an independent expert panel of clinicians. Follow-up will continue in the longer term, including through electronic health record linkage.

Value: To our knowledge, the study is the first to assess the clinical value of invasive management guided by routine use of adjunctive tests of coronary function in appropriately selected patients. The study will provide new insights into disease mechanisms and provide pilot data to inform the rationale and design of a larger clinical trial. The CMR substudy will provide information on the diagnostic utility of quantitative non-invasive imaging methods in this patient population. Should our hypotheses be confirmed, the research will bring new knowledge with potential benefits to patients and healthcare providers.

ELIGIBILITY:
Inclusion Criteria:

A clinically-indicated plan for invasive coronary angiography. Symptoms of angina or angina-equivalent (according to the Rose- and Seattle Angina questionnaires).

Exclusion Criteria:

A non-coronary indication for invasive angiography e.g. valve disease During the angiogram: obstructive disease evident in a main coronary artery (diameter >2.5 mm), i.e. a coronary stenosis>50% or a fractional flow reserve (FFR) ≤0.80 Lack of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2016-11-07 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-11-06 (Actual)

PRIMARY OUTCOMES:
Health status (Seattle Angina Score) | 6 months
  Health status and symptoms will be assessed at baseline and again at 6 months using the Seattle Angina Questionnaire. The primary outcome is the within-subject change in SAQ score at 6 months from baseline.

SECONDARY OUTCOMES:
Feasibility of the stratified medicine approach defined by protocol compliance as measured by deviations from the protocol. | Through study completion, 3 years
  Feasibility will be assessed in terms of enrolment rates and protocol compliance relating to enrolment, cross-over, integrity of blinding, adherence with therapy during follow-up, and compliance with follow up assessments
Procedure-related serious adverse events | Day 1 (index coronary angiogram procedure)
  Safety as reflected by the occurrence of procedure-related serious adverse events
Prevalence of endotypes | Day 1
  Diagnosis of endotypes (disease strata): obstructive CAD, coronary vasospastic angina, microvascular angina, endothelial dysfunction (no angina), normal (non-cardiac, normal coronary function results, no angina).
Diagnostic utility of the diagnostic intervention | Day 1
  Impact of disclosure of the coronary function test results on the diagnosis and certainty of the diagnosis (diagnostic utility)
Clinical utility of the stratified approach | Day 1
  Impact of disclosure of the coronary function test results on medical decisions (including treatment and investigations), and to compare these decisions against a medical decisions formed by an independent panel of experts (reference dataset)
Cardiovascular risk factors | Day 1
  Assess the relationships between cardiovascular risk factors, reflected by validated risk scores (e.g. ASSIGN, JBS3), and parameters of coronary function, in medically managed patients.
Anxiety and depression | Through study completion, 3 years
  Assess the participants' self-reported levels of anxiety and depression using the Patient Health Questionnaire-4 (PHQ-4)
Treatment satisfaction | Through study completion, 3 years
  Assess the participants' self-reported levels of treatment satisfaction using the Treatment Satisfaction Questionnaire for Medication (TSQM)
Illness perception | Through study completion, 3 years
  Assess the participants' perception of their illness using the brief Illness Perception Questionnaire
Health status EQ5D | Through study completion, 3 years
  Assess the participants' general health status and self reported quality of life using the EQ5D questionnaire.
Health status (Seattle Angina Score) | Through study completion, 3 years
  Health status and symptoms will be assessed at baseline and again at 6 months, 12 months and close-out using the Seattle Angina Questionnaire. The secondary outcome is the within-subject change in SAQ score over time.
Biomarkers | 36 months
  Assess associations between circulating molecules that are implicated in the pathophysiology of disorders of coronary function.
Health economics | 36 months
  Assess resource utilisation including primary and secondary care costs for tests, procedures and out-patient visits, and medicines, between the randomised groups
Myocardial perfusion | 42 days
  Assess the diagnostic accuracy of stress perfusion magnetic resonance imaging for identification of endotypes based on reference tests of coronary function.
Incidental findings | 42 days
  Detection of clinically significant (actionable) incidental findings using magnetic resonance imaging. The incidental findings may be cardiac or non-cardiac.
Myocardial tissue characterisation | 42 days
  Detection of myocardial pathology using multiparametric CMR

CONTACTS AND LOCATIONS:
Overall Officials: Katriona Brooksbank, PhD, Study Director — University of Glasgow
Locations (2):
- United Kingdom (2):
  - Golden Jubilee National Hospital, Clydebank, Dunbartonshire
  - Hairmyres Hospital, East Kilbride, Lanarkshire

IPD SHARING:
Plan to Share IPD: Undecided
Data access may be possible pending Sponsor approval

REFERENCES:
- [Background] Ford TJ, Ong P, Sechtem U, Beltrame J, Camici PG, Crea F, Kaski JC, Bairey Merz CN, Pepine CJ, Shimokawa H, Berry C; COVADIS Study Group. Assessment of Vascular Dysfunction in Patients Without Obstructive Coronary Artery Disease: Why, How, and When. JACC Cardiovasc Interv. 2020 Aug 24;13(16):1847-1864. doi: 10.1016/j.jcin.2020.05.052. PMID 32819476
- [Background] Ford TJ, Corcoran D, Sidik N, Oldroyd KG, Rocchiccioli P, McEntegart M, Berry C. MINOCA: Requirement for Definitive Diagnostic Work-Up. Heart Lung Circ. 2019 Feb;28(2):e4-e6. doi: 10.1016/j.hlc.2018.04.001. No abstract available. PMID 30654950
- [Background] Collison D, Copt S, Mizukami T, Collet C, McLaren R, Didagelos M, Aetesam-Ur-Rahman M, McCartney P, Ford TJ, Lindsay M, Shaukat A, Rocchiccioli P, Brogan R, Watkins S, McEntegart M, Good R, Robertson K, O'Boyle P, Davie A, Khan A, Hood S, Eteiba H, Berry C, Oldroyd KG. Angina After Percutaneous Coronary Intervention: Patient and Procedural Predictors. Circ Cardiovasc Interv. 2023 Apr;16(4):e012511. doi: 10.1161/CIRCINTERVENTIONS.122.012511. Epub 2023 Mar 28. PMID 36974680
- [Background] Rush CJ, Berry C, Oldroyd KG, Rocchiccioli JP, Lindsay MM, Touyz RM, Murphy CL, Ford TJ, Sidik N, McEntegart MB, Lang NN, Jhund PS, Campbell RT, McMurray JJV, Petrie MC. Prevalence of Coronary Artery Disease and Coronary Microvascular Dysfunction in Patients With Heart Failure With Preserved Ejection Fraction. JAMA Cardiol. 2021 Oct 1;6(10):1130-1143. doi: 10.1001/jamacardio.2021.1825. PMID 34160566
- [Background] Kunadian V, Chieffo A, Camici PG, Berry C, Escaned J, Maas AHEM, Prescott E, Karam N, Appelman Y, Fraccaro C, Louise Buchanan G, Manzo-Silberman S, Al-Lamee R, Regar E, Lansky A, Abbott JD, Badimon L, Duncker DJ, Mehran R, Capodanno D, Baumbach A. An EAPCI Expert Consensus Document on Ischaemia with Non-Obstructive Coronary Arteries in Collaboration with European Society of Cardiology Working Group on Coronary Pathophysiology & Microcirculation Endorsed by Coronary Vasomotor Disorders International Study Group. Eur Heart J. 2020 Oct 1;41(37):3504-3520. doi: 10.1093/eurheartj/ehaa503. PMID 32626906
- [Background] Vrints C, Andreotti F, Koskinas KC, Rossello X, Adamo M, Ainslie J, Banning AP, Budaj A, Buechel RR, Chiariello GA, Chieffo A, Christodorescu RM, Deaton C, Doenst T, Jones HW, Kunadian V, Mehilli J, Milojevic M, Piek JJ, Pugliese F, Rubboli A, Semb AG, Senior R, Ten Berg JM, Van Belle E, Van Craenenbroeck EM, Vidal-Perez R, Winther S; ESC Scientific Document Group. 2024 ESC Guidelines for the management of chronic coronary syndromes. Eur Heart J. 2024 Sep 29;45(36):3415-3537. doi: 10.1093/eurheartj/ehae177. No abstract available. PMID 39210710
- [Background] Cannon RO 3rd, Leon MB, Watson RM, Rosing DR, Epstein SE. Chest pain and "normal" coronary arteries--role of small coronary arteries. Am J Cardiol. 1985 Jan 25;55(3):50B-60B. doi: 10.1016/0002-9149(85)90613-7. PMID 3969858
- [Background] Cannon RO 3rd, Bonow RO, Bacharach SL, Green MV, Rosing DR, Leon MB, Watson RM, Epstein SE. Left ventricular dysfunction in patients with angina pectoris, normal epicardial coronary arteries, and abnormal vasodilator reserve. Circulation. 1985 Feb;71(2):218-26. doi: 10.1161/01.cir.71.2.218. PMID 3965167
- [Background] Sax FL, Cannon RO 3rd, Hanson C, Epstein SE. Impaired forearm vasodilator reserve in patients with microvascular angina. Evidence of a generalized disorder of vascular function? N Engl J Med. 1987 Nov 26;317(22):1366-70. doi: 10.1056/NEJM198711263172202. PMID 3683470
- [Background] Kaski JC, Elliott PM, Salomone O, Dickinson K, Gordon D, Hann C, Holt DW. Concentration of circulating plasma endothelin in patients with angina and normal coronary angiograms. Br Heart J. 1995 Dec;74(6):620-4. doi: 10.1136/hrt.74.6.620. PMID 8541166
- [Background] Elliott PM, Krzyzowska-Dickinson K, Calvino R, Hann C, Kaski JC. Effect of oral aminophylline in patients with angina and normal coronary arteriograms (cardiac syndrome X). Heart. 1997 Jun;77(6):523-6. doi: 10.1136/hrt.77.6.523. PMID 9227295
- [Background] Beltrame JF, Crea F, Kaski JC, Ogawa H, Ong P, Sechtem U, Shimokawa H, Bairey Merz CN; Coronary Vasomotion Disorders International Study Group (COVADIS). The Who, What, Why, When, How and Where of Vasospastic Angina. Circ J. 2016;80(2):289-98. doi: 10.1253/circj.CJ-15-1202. Epub 2015 Dec 18. PMID 26686994
- [Background] Williams MC, Hunter A, Shah A, Assi V, Lewis S, Mangion K, Berry C, Boon NA, Clark E, Flather M, Forbes J, McLean S, Roditi G, van Beek EJ, Timmis AD, Newby DE; Scottish COmputed Tomography of the HEART (SCOT-HEART) Trial Investigators. Symptoms and quality of life in patients with suspected angina undergoing CT coronary angiography: a randomised controlled trial. Heart. 2017 Jul;103(13):995-1001. doi: 10.1136/heartjnl-2016-310129. Epub 2017 Feb 28. PMID 28246175
- [Background] Ford TJ, Corcoran D, Berry C. Coronary artery disease: physiology and prognosis. Eur Heart J. 2017 Jul 1;38(25):1990-1992. doi: 10.1093/eurheartj/ehx226. No abstract available. PMID 28549103
- [Background] Ford TJ, Berry C. Angina: contemporary diagnosis and management. Heart. 2020 Mar;106(5):387-398. doi: 10.1136/heartjnl-2018-314661. Epub 2020 Feb 12. No abstract available. PMID 32054665
- [Background] Sidik NP, McEntegart M, Roditi G, Ford TJ, McDermott M, Morrow A, Byrne J, Adams J, Hargreaves A, Oldroyd KG, Stobo D, Wu O, Messow CM, McConnachie A, Berry C. Rationale and design of the British Heart Foundation (BHF) Coronary Microvascular Function and CT Coronary Angiogram (CorCTCA) study. Am Heart J. 2020 Mar;221:48-59. doi: 10.1016/j.ahj.2019.11.015. Epub 2019 Dec 2. PMID 31911341
- [Background] Ford TJ, Yii E, Sidik N, Good R, Rocchiccioli P, McEntegart M, Watkins S, Eteiba H, Shaukat A, Lindsay M, Robertson K, Hood S, McGeoch R, McDade R, McCartney P, Corcoran D, Collison D, Rush C, Stanley B, McConnachie A, Sattar N, Touyz RM, Oldroyd KG, Berry C. Ischemia and No Obstructive Coronary Artery Disease: Prevalence and Correlates of Coronary Vasomotion Disorders. Circ Cardiovasc Interv. 2019 Dec;12(12):e008126. doi: 10.1161/CIRCINTERVENTIONS.119.008126. Epub 2019 Dec 13. PMID 31833416
- [Background] Ford TJ, Stanley B, Sidik N, Good R, Rocchiccioli P, McEntegart M, Watkins S, Eteiba H, Shaukat A, Lindsay M, Robertson K, Hood S, McGeoch R, McDade R, Yii E, McCartney P, Corcoran D, Collison D, Rush C, Sattar N, McConnachie A, Touyz RM, Oldroyd KG, Berry C. 1-Year Outcomes of Angina Management Guided by Invasive Coronary Function Testing (CorMicA). JACC Cardiovasc Interv. 2020 Jan 13;13(1):33-45. doi: 10.1016/j.jcin.2019.11.001. Epub 2019 Nov 11. PMID 31709984
- [Background] Ford TJ, Berry C. How to Diagnose and Manage Angina Without Obstructive Coronary Artery Disease: Lessons from the British Heart Foundation CorMicA Trial. Interv Cardiol. 2019 May 21;14(2):76-82. doi: 10.15420/icr.2019.04.R1. eCollection 2019 May. PMID 31178933
- [Background] Corcoran D, Ford TJ, Hsu LY, Chiribiri A, Orchard V, Mangion K, McEntegart M, Rocchiccioli P, Watkins S, Good R, Brooksbank K, Padmanabhan S, Sattar N, McConnachie A, Oldroyd KG, Touyz RM, Arai A, Berry C. Rationale and design of the Coronary Microvascular Angina Cardiac Magnetic Resonance Imaging (CorCMR) diagnostic study: the CorMicA CMR sub-study. Open Heart. 2018 Dec 30;5(2):e000924. doi: 10.1136/openhrt-2018-000924. eCollection 2018. PMID 30687508
- [Background] Ford TJ, Rocchiccioli P, Good R, McEntegart M, Eteiba H, Watkins S, Shaukat A, Lindsay M, Robertson K, Hood S, Yii E, Sidik N, Harvey A, Montezano AC, Beattie E, Haddow L, Oldroyd KG, Touyz RM, Berry C. Systemic microvascular dysfunction in microvascular and vasospastic angina. Eur Heart J. 2018 Dec 7;39(46):4086-4097. doi: 10.1093/eurheartj/ehy529. PMID 30165438
- [Derived] Ford TJ, Corcoran D, Padmanabhan S, Aman A, Rocchiccioli P, Good R, McEntegart M, Maguire JJ, Watkins S, Eteiba H, Shaukat A, Lindsay M, Robertson K, Hood S, McGeoch R, McDade R, Yii E, Sattar N, Hsu LY, Arai AE, Oldroyd KG, Touyz RM, Davenport AP, Berry C. Genetic dysregulation of endothelin-1 is implicated in coronary microvascular dysfunction. Eur Heart J. 2020 Sep 7;41(34):3239-3252. doi: 10.1093/eurheartj/ehz915. PMID 31972008
- [Derived] Ford TJ, Stanley B, Good R, Rocchiccioli P, McEntegart M, Watkins S, Eteiba H, Shaukat A, Lindsay M, Robertson K, Hood S, McGeoch R, McDade R, Yii E, Sidik N, McCartney P, Corcoran D, Collison D, Rush C, McConnachie A, Touyz RM, Oldroyd KG, Berry C. Stratified Medical Therapy Using Invasive Coronary Function Testing in Angina: The CorMicA Trial. J Am Coll Cardiol. 2018 Dec 11;72(23 Pt A):2841-2855. doi: 10.1016/j.jacc.2018.09.006. Epub 2018 Sep 25. PMID 30266608
- See also: Cardiology and Imaging Group, University of Glasgow — https://www.gla.ac.uk/researchinstitutes/icams/staff/colinberry
- See also: British Heart Foundation — https://www.bhf.org.uk/research